CLINICAL TRIAL: NCT02532621
Title: Clinical Evaluation of a Vascular Venous Anastomotic Connector for Minimally Invasive Connection of an Arteriovenous Graft for Hemodialysis [InterGraft VIG-only Study]
Brief Title: Clinical Evaluation of a Vascular Venous Anastomotic Connector [InterGraft VIG-only Study]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phraxis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Venous Anastomotic Connector
Record Dates: First submitted 2015-08-19; First posted 2015-08-26 (Estimated); Results first posted 2025-01-01 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Venous InterGraft Connector (VIG) (Experimental): This is a nonrandomized, single-arm study: All enrolled patients are assigned to the same treatment: AVG implantation using a VIG (study device) to create the venous anastomosis and standard suturing to create the arterial anastomosis of the implanted AVG.
  Interventions: Device: Venous InterGraft Connector; Procedure: sutured arterial anastomosis of an implanted vascular graft for hemodialysis; Procedure: hemodialysis

INTERVENTIONS:
Device: Venous InterGraft Connector — The device is designed for transcatheter delivery within a vein and connection to an AVG that has been tunneled under the skin in a standard manner. The connection is made via a small skin incision.
  Other Names: VIG
Procedure: sutured arterial anastomosis of an implanted vascular graft for hemodialysis — The arterial anastomosis of the implanted vascular graft for hemodialysis is formed using standard suturing technique.
Procedure: hemodialysis — The implanted vascular graft is intended as a vascular access for performing hemodialysis treatments.

SUMMARY:
The InterGraft™ Venous Anastomotic Connector provides an endovascular, minimally invasive means for attachment of an arteriovenous graft to a vein in the upper extremity. The InterGraft™ Venous Anastomotic Connector facilitates creation of the arteriovenous graft connection to a vein in support of hemodialysis in subjects with End Stage Renal Disease. The InterGraft™ Venous Anastomotic Connector is used together with conventional suturing of the arterial anastomosis to facilitate creation of an arteriovenous graft in support of hemodialysis in subjects with End Stage Renal Disease.

DETAILED DESCRIPTION:
The InterGraft™ Venous Anastomotic Connector (VIG) was developed for endovascular, minimally invasive venous anastomosis of a standard arteriovenous graft (AVG) for hemodialysis. This study will evaluate the safety and performance of the VIG for anastomosis of a commercially available, 6 mm diameter, synthetic AVG. Anastomoses with the VIG may potentially reduce venous vessel trauma, improve the local vessel wall shear stresses and promote laminar flow, thereby improving patency.

While recognizing that a native fistula is the recommended access for hemodialysis, AVGs remain a frequently used access type. This study focuses on subjects who have a failed fistula, cannot have a fistula or are better suited for an AVG, as determined by the physician. The implant procedural outcomes, the number and type of major adverse events, and patency throughout a six-month follow-up period will be evaluated. The six-month patency rate will be compared with a pre-specified patency performance goal drawn from surgical AVG literature and published performance standards.

This is a pivotal, multicenter, prospective, non-randomized design study. All enrolled subjects will receive the VIG device and will have a standard sutured arterial anastomosis.

A total of 158 evaluable subjects will be enrolled, defined as primary analysis population of 146 subjects plus allowance for 12 subjects lost-to-follow up.

The study includes10 participating clinical centers. Study site investigators are physicians skilled in AVG placement and interventional techniques. Study data will be collected up to the point at which each subject has completed the six-month endpoint or experienced a terminal study endpoint.

The study will be conducted in compliance with the Investigational Plan, Investigational Device Exemption regulations, Good Clinical Practice guidelines, and other applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age.
2. Subject requires the creation of a vascular access graft for hemodialysis, secondary to a diagnosis of End Stage Renal Disease.
3. Subject is able to have the vascular access graft placed in an upper extremity.
4. Baseline imaging shows suitable vascular anatomy/ vessel size for the InterGraft™ Venous Connector and an artery at least 3.5 mm in diameter that is suitable for creating the arterial anastomosis.
5. Subject has a reasonable expectation of remaining on hemodialysis for at least 6 months.
6. Subject or his/her legal guardian understands the study and is willing and able to comply with the dialysis schedule and follow-up requirements.
7. Subject or his/her legal guardian provides written informed consent. NOTE: In accordance with the requirements of some Institutional Review Boards, where applicable, only those subjects with capacity to consent for themselves will be included. Thus, where required by the Institutional Review Board, adult individuals who lack capacity to consent for themselves will be excluded from the study.
8. Physician's examination at time of surgery shows no significant vessel lesions, calcification(s), anatomic structures or abnormalities that may limit ability to safely deploy the InterGraft Connectors or create a sutured arterial anastomosis.

Exclusion Criteria:

1. Subject has a documented and unsuccessfully treated ipsilateral central venous stenosis as determined by imaging.
2. Subject currently has a known or suspected bacterial, fungal, or HIV infection. NOTE: Patients with hepatitis B or C may be included in the study.
3. Subject has a known hypercoagulable or bleeding disorder or requires treatment with warfarin or heparin.

   NOTE: The intent of this criterion is to exclude patients with high risk for bleeding or clotting complications. As such, patients who are taking oral anticoagulants (blood thinners) including, but not limited to, Xarelto® (rivaroxaban) or Eliquis® (apixaban) should also be excluded from the study. Patients may receive anticoagulation therapy any time after the study AV graft implant procedure, at their physician's discretion. This should be driven by an indication unrelated to the vascular access.
4. Subject has had a previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or has known sensitivity to heparin.
5. Subject has co-morbid conditions that may limit their ability to comply with study and follow-up requirements.
6. The patient has had >2 previous arteriovenous accesses in treatment arm.
7. Subject is currently taking Aggrenox®.
8. Subject is in need of, or is scheduled for any major surgery within 30 days of the study procedure.
9. Subject is currently taking maintenance immunosuppressant medication such as rapamycin, mycophenolate or mycophenolic acid, prednisone (>10 mg), cyclosporine, tacrolimus or cyclophosphamide.
10. Life expectancy is less than 12 months.
11. Subject is pregnant. NOTE: A negative urine pregnancy test within 24 hours of the study procedure is required in all female subjects with reproductive capacity.
12. Subject is a poor compliance risk (i.e. history of IV or oral drug abuse).
13. The subject is enrolled in another dialysis or vascular investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy M Setum, Ph.D, Study Director — Phraxis, Inc.; John R Ross, M.D., Principal Investigator — Regional Medical Center
Locations (10):
- United States (10):
  - Triad of Alabama/Flowers Hospital, Dothan, Alabama
  - Cartersville Medical Center, LLC, Cartersville, Georgia
  - Medical Center of Central Georgia - Navicent Health, Macon, Georgia
  - Henry Ford Health System- Dept of Surgery, Detroit, Michigan
  - Saint Louis University, St Louis, Missouri
  - Surgical Specialists of Charlotte, Charlotte, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Physician Associates II, Florence, South Carolina
  - Regional Medical Center of Orangeburg and Calhoun Counties, Orangeburg, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Renal Data System. USRDS 2011 Annual Data Report: Volume 2. Atlas of End Stage Renal Disease in the United States. Bethesda, MD, National Institutes of Health, National Institutes of Diabetes, and Digestive and Kidney Diseases; 2011
- [Background] Dember LM, Beck GJ, Allon M, Delmez JA, Dixon BS, Greenberg A, Himmelfarb J, Vazquez MA, Gassman JJ, Greene T, Radeva MK, Braden GL, Ikizler TA, Rocco MV, Davidson IJ, Kaufman JS, Meyers CM, Kusek JW, Feldman HI; Dialysis Access Consortium Study Group. Effect of clopidogrel on early failure of arteriovenous fistulas for hemodialysis: a randomized controlled trial. JAMA. 2008 May 14;299(18):2164-71. doi: 10.1001/jama.299.18.2164. PMID 18477783
- [Background] Akoh JA. Prosthetic arteriovenous grafts for hemodialysis. J Vasc Access. 2009 Jul-Sep;10(3):137-47. doi: 10.1177/112972980901000301. PMID 19670164
- [Background] Roy-Chaudhury P, Kelly BS, Zhang J, Narayana A, Desai P, Melham M, Duncan H, Heffelfinger SC. Hemodialysis vascular access dysfunction: from pathophysiology to novel therapies. Blood Purif. 2003;21(1):99-110. doi: 10.1159/000067863. PMID 12596755
- [Background] Lee T, Roy-Chaudhury P. Advances and new frontiers in the pathophysiology of venous neointimal hyperplasia and dialysis access stenosis. Adv Chronic Kidney Dis. 2009 Sep;16(5):329-38. doi: 10.1053/j.ackd.2009.06.009. PMID 19695501
- [Background] Lok CE, Allon M, Moist L, Oliver MJ, Shah H, Zimmerman D. Risk equation determining unsuccessful cannulation events and failure to maturation in arteriovenous fistulas (REDUCE FTM I). J Am Soc Nephrol. 2006 Nov;17(11):3204-12. doi: 10.1681/ASN.2006030190. Epub 2006 Sep 20. PMID 16988062
- [Background] Lee HW, Allon M. When should a patient receive an arteriovenous graft rather than a fistula? Semin Dial. 2013 Jan-Feb;26(1):6-10. doi: 10.1111/sdi.12040. Epub 2012 Nov 22. PMID 23173947
- [Background] Saran R, Robinson B, Abbott KC, Agodoa LY, Albertus P, Ayanian J, Balkrishnan R, Bragg-Gresham J, Cao J, Chen JL, Cope E, Dharmarajan S, Dietrich X, Eckard A, Eggers PW, Gaber C, Gillen D, Gipson D, Gu H, Hailpern SM, Hall YN, Han Y, He K, Hebert H, Helmuth M, Herman W, Heung M, Hutton D, Jacobsen SJ, Ji N, Jin Y, Kalantar-Zadeh K, Kapke A, Katz R, Kovesdy CP, Kurtz V, Lavalee D, Li Y, Lu Y, McCullough K, Molnar MZ, Montez-Rath M, Morgenstern H, Mu Q, Mukhopadhyay P, Nallamothu B, Nguyen DV, Norris KC, O'Hare AM, Obi Y, Pearson J, Pisoni R, Plattner B, Port FK, Potukuchi P, Rao P, Ratkowiak K, Ravel V, Ray D, Rhee CM, Schaubel DE, Selewski DT, Shaw S, Shi J, Shieu M, Sim JJ, Song P, Soohoo M, Steffick D, Streja E, Tamura MK, Tentori F, Tilea A, Tong L, Turf M, Wang D, Wang M, Woodside K, Wyncott A, Xin X, Zang W, Zepel L, Zhang S, Zho H, Hirth RA, Shahinian V. US Renal Data System 2016 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2017 Mar;69(3 Suppl 1):A7-A8. doi: 10.1053/j.ajkd.2016.12.004. No abstract available. PMID 28236831
- [Result] Burgess JS, Beaver JD, London M, Rohan V, Orland P, Yevzlin A, Setum C, Ross J; InterGraft Study Investigators. Prospective multicenter study of a novel endovascular venous anastomotic procedure and device for implantation of an arteriovenous graft for hemodialysis. J Vasc Access. 2024 Jul;25(4):1244-1251. doi: 10.1177/11297298231159691. Epub 2023 Mar 9. PMID 36895157

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Venous InterGraft Connector (VIG)
Started | 158
Completed | 132
Not Completed | 26
Not completed — Death | 3
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 6
Not completed — implanted graft abandoned before 6 months | 12
Not completed — last follow up performed outside window (<166 days) -censored | 2

BASELINE CHARACTERISTICS:
Arm/Group | Venous InterGraft Connector (VIG)
Number analyzed (Participants) | 158
Age, Continuous [Mean (Full Range); unit: years] | 62.6 [24.0 to 92.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 154
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 123
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Diabetes mellitus [Count of Participants; unit: Participants] | 98
Obesity [Count of Participants; unit: Participants] | 51
Hypertension [Count of Participants; unit: Participants] | 89
Cardiovascular Disease [Count of Participants; unit: Participants] | 78
Number of prior permanent vascular access(s) for hemodialysis [Count of Participants; unit: Participants]
  0 | 64
  1 | 66
  2 or more | 28
Duration of Hemodialysis [Count of Participants; unit: Participants]
  < 6 months | 69
  >= 6 months and <12 months | 15
  >= 12 months | 59
  NA (no current hemodialysis) | 15
Current hemodialysis using a catheter [Count of Participants; unit: Participants] | 134

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Patency at 6 Months
Description: Percentage of subjects free from loss of access of the study graft for hemodialysis
Time Frame: Six months of clinical follow-up following treatment assignment (enrollment)
Population: Intention-to-treat analysis population (All patients assigned to treatment using the study device). Patients withdrawn for reasons other than loss of cumulative patency were included in the analysis up until the time of withdrawal and were considered censored in the analysis, after withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Venous InterGraft Connector (VIG)
Number analyzed (Participants) | 158
Participants | 146
Statistical Analysis 1: Comparison: Venous InterGraft Connector (VIG); The primary endpoint was evaluated by comparison with a performance goal of 75% that was determined from medical literature. The sample size of 158 patients was estimated as follows: * Kaplan-Meier estimate of cumulative patency rate at 6 months (exact binomial estimation for sample size) * Type I error (alpha): 0.025 (one-sided) * 80% Statistical power * 8% Lost-to-follow up rate; Test type: Non-Inferiority — Cumulative patency at 6 months was evaluated using the estimated patency from a Kaplan Meier survival analysis. The test statistic took the following form: Z-test statistic = (P - 0.75) / SE (P) Where, (P) represents the Kaplan Meier estimate of cumulative patency at 6 months, and the standard error SE (P) is estimated using the method of Peto et al (1977); p < 0.001, one-sided binomial exact test — A one-sided p-value of 0.025 was considered evidence of statistical significance for the primary study endpoint; Cumulative patency = 92.1

2. Secondary Outcome: Acute Device Success
Description: AV graft flow at end of implant procedure
Time Frame: 24 hours
Population: Intention-to-treat (all patients assigned to treatment using the study device)
Measure: Count of Participants; unit: Participants
Arm/Group | Venous InterGraft Connector (VIG)
Number analyzed (Participants) | 158
Participants | 158

3. Secondary Outcome: Primary Unassisted Patency
Description: Percentage of subjects free from the occurrence of either access thrombosis or an access procedure performed to maintain access patency
Time Frame: Six months
Population: Intention-to-treat (all patients assigned to treatment using the study device). Patients withdrawn for reasons other than loss of primary unassisted patency were included in the analysis up until the time of withdrawal and were considered censored in the analysis, according to usual convention, after withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Venous InterGraft Connector (VIG)
Number analyzed (Participants) | 158
Participants | 95

4. Secondary Outcome: Time to First Cannulation
Description: Time from initial access placement to first graft cannulation for hemodialysis
Time Frame: Six months
Population: Intention-to-treat.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Venous InterGraft Connector (VIG)
Number analyzed (Participants) | 158
days | 20.1 (23.5)

5. Secondary Outcome: Interventions Required to Maintain Patency
Description: Number of interventions required to maintain secondary patency
Time Frame: Six months
Population: intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Venous InterGraft Connector (VIG)
Number analyzed (Participants) | 158
Participants
  One intervention to maintain AVG patency | 33
  Two interventions to maintain AVF patency | 14
  Three or more interventions to maintain AVG patency | 8
  No interventions to maintain AVG patency | 103

6. Secondary Outcome: Serious Adverse Events (Secondary Endpoint Defined SAEs)
Description: Number and type of serious adverse events- death, emergent surgery, significant bleeding,graft infection, pseudoaneurysm
Time Frame: Six months
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Venous InterGraft Connector (VIG)
Number analyzed (Participants) | 158
Participants
  Death | 3
  AVG infection | 6
  significant bleeding | 0
  emergent surgery | 0
  pseudoaneurysm | 0
  No protocol-defined SAEs | 149

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the date of enrollment (date of index procedure) through 6 months or until the occurrence of a terminal study event (death, lost to follow up, withdrew from the study, abandonment of implanted graft), whichever occurred first.
Description: Serious adverse events were to be initially reported to the Sponsor within 24 hours of discovery by the investigator.
Arm/Group | Venous InterGraft Connector (VIG)
All-Cause Mortality (participants affected / at risk) | 3/158
Serious Adverse Events (participants affected / at risk) | 58/158
Other Adverse Events (participants affected / at risk) | 37/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venous InterGraft Connector (VIG) (N=158)
graft/access circuit infection (Infections and infestations) | 6 (6) — Graft infection is a protocol-specified SAE (secondary endpoint)
Emergent surgery (Surgical and medical procedures) | 0 (0) — Emergent surgery is a protocol-specified SAE (secondary endpoint)
Significant bleeding (Vascular disorders) | 0 (0) — Significant bleeding is a protocol-specified SAE (secondary endpoint)
Pseudoaneurysm (Vascular disorders) | 0 (0) — Pseudoaneurysm is a protocol-specified SAE (secondary endpoint)
sepsis (Infections and infestations) | 4 (4)
cellulitis (Infections and infestations) | 2 (2)
Abscess, general (Infections and infestations) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
gangrene (Infections and infestations) | 1 (1)
other infection (not AVG) (Infections and infestations) | 1 (1)
intervertebral discitis (Infections and infestations) | 1 (1)
sinusitis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
urosepsis (Infections and infestations) | 1 (1)
death (General disorders) | 2 (2)
pyrexia (General disorders) | 2 (2)
asthenia (General disorders) | 1 (1)
hemorrhage, catheter site (General disorders) | 1 (1)
chest discomfort (General disorders) | 1 (1)
chest pain (General disorders) | 1 (1)
peripheral swelling (General disorders) | 1 (1)
stent malfunction (General disorders) | 1 (1)
acute myocardial infarction (Cardiac disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1)
cardiac failure (Cardiac disorders) | 1 (1)
cardiac failure, acute (Cardiac disorders) | 1 (1)
cardiac failure, chronic (Cardiac disorders) | 1 (1)
cardiac failure, congestive (Cardiac disorders) | 1 (1)
cardio-respiratory arrest (Cardiac disorders) | 1 (1)
coronary artery disease (Cardiac disorders) | 1 (1)
steal syndrome (Vascular disorders) | 4 (6)
hypertensive emergency (Vascular disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
ischemia (Vascular disorders) | 1 (1)
malignant hypertension (Vascular disorders) | 1 (1)
fluid overload (Metabolism and nutrition disorders) | 2 (2)
hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
failure to thrive (Metabolism and nutrition disorders) | 1 (1)
cerebral hemorrhage (Nervous system disorders) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 1 (1)
Diziness (Nervous system disorders) | 1 (1)
embolic stroke (Nervous system disorders) | 1 (1)
encephalopathy (Nervous system disorders) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1)
GI hemorrhage (Gastrointestinal disorders) | 1 (1)
impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
intestinal ischemia (Gastrointestinal disorders) | 1 (1)
melena (Gastrointestinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
blood pressure management (Surgical and medical procedures) | 1 (1)
hospitalization, general (Surgical and medical procedures) | 1 (1)
parathyroidectomy (Surgical and medical procedures) | 1 (1)
amputation, toe (Surgical and medical procedures) | 1 (1)
pain, procedure (Injury, poisoning and procedural complications) | 1 (1)
vascular graft complication (Injury, poisoning and procedural complications) | 1 (1)
fracture, wrist (Injury, poisoning and procedural complications) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 1 (1)
hematuria (Renal and urinary disorders) | 1 (1)
urinary retention (Renal and urinary disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 2 (2)
hepatic failure (Hepatobiliary disorders) | 1 (1)
heart rate decrease (Investigations) | 1 (1)
pain, extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
mental status change (Psychiatric disorders) | 1 (1)
facial swelling (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venous InterGraft Connector (VIG) (N=158)
swelling, implant site (General disorders) | 8 (8)
chest pain (General disorders) | 1 (1)
pain, implant site (General disorders) | 1 (1)
pyrexia (General disorders) | 1 (1)
pain, suprapubic (General disorders) | 1 (1)
vascular steal syndrome (Vascular disorders) | 8 (8)
hemorrhage (Vascular disorders) | 2 (2)
diabetic microangiopathy (Vascular disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (2)
coldness, peripheral (Vascular disorders) | 1 (1)
contusion (Injury, poisoning and procedural complications) | 3 (4)
graft complication (Injury, poisoning and procedural complications) | 2 (2)
AV site complication (Injury, poisoning and procedural complications) | 1 (1)
fracture (Injury, poisoning and procedural complications) | 1 (1)
incision site vesicles (Injury, poisoning and procedural complications) | 1 (1)
hemorrhage, post procedure (not serious) (Injury, poisoning and procedural complications) | 1 (1)
seroma (Injury, poisoning and procedural complications) | 1 (1)
pseudoaneurysm (not requiring treatment) (Injury, poisoning and procedural complications) | 1 (1)
hypoasthesia (Nervous system disorders) | 2 (2)
neuralgia (Nervous system disorders) | 2 (2)
paresthesia (Nervous system disorders) | 2 (2)
diziness (Nervous system disorders) | 1 (2)
sciatica (Nervous system disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 2 (2)
colitis, microscopic (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
erythema (Skin and subcutaneous tissue disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
conjunctivitis (Infections and infestations) | 1 (1)
infection, minor (Infections and infestations) | 1 (1)
diverticulitis (Infections and infestations) | 1 (1)
decreased appetite (Metabolism and nutrition disorders) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
pain, extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
stiffness, musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
ER examination (Investigations) | 1 (1)
breast pain (Reproductive system and breast disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study had the usual limitations associated with a non-randomized investigation, and this was mitigated by use of the robust historical literature to define the 6-month patency PG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results proposed to be published or presented shall be submitted to Sponsor for review and comment at least 45 days prior to submission to allow Sponsor to protect its rights to any patentable inventions disclosed and to permit Sponsor to request removal of any Confidential Information provided by Sponsor.

Any such publication or presentation shall acknowledge, as appropriate, the contribution of Sponsor, its employees, agents and representatives.

DOCUMENTS (2):
  • Study Protocol (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT02532621/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT02532621/SAP_001.pdf